CLINICAL TRIAL: NCT00186628
Title: An Open-label, Phase 2 Trial of Prophylactic Rituximab Therapy for Prevention of Chronic Graft Versus Host Disease After TLI/ARG Nonmyeloablative Allogeneic Stem Cell Transplantation
Brief Title: Phase 2 Trial of Prophylactic Rituximab Therapy for Prevention of CGVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Miklos, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-02372; 96160 (Other: Stanford Secondary IRB Approval Number); BMT172 (Other: OnCore); SPO (Other: Leukemia & Lymphoma Society); P01CA049605 (NIH); NCT00234013 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Leukemia, Mast-Cell; Mantle-cell Lymphoma
MeSH Terms: conditions — Leukemia, Mast-Cell; Lymphoma, Mantle-Cell | interventions — Rituximab; thymoglobulin; Cyclosporine; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor; Granisetron; Methylprednisolone Hemisuccinate; Methylprednisolone; Methylprednisolone Acetate; Acetaminophen; Diphenhydramine; Hydrocortisone; hydrocortisone valerate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prophylactic Rituximab (Experimental): Rituximab will be infused after a non-myeloablative transplantation regimen of total lymphoid irradiation (TLI) + anti-thymoglobulin (ATG), with the intention of reducing chronic graft-vs-host disease (cGvHD)
  Interventions: Procedure: Total lymphoid irradiation; Drug: Rituximab; Drug: Anti-thymoglobulin, rabbit (ATG, rabbit ATG); Drug: Cyclosporine; Drug: Mycophenylate mofetil; Drug: Filgrastim; Drug: Granisetron; Drug: Solumedrol; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Hydrocortisone

INTERVENTIONS:
Procedure: Total lymphoid irradiation — Total lymphoid irradiation (TLI) administered at 80cGy for 10 days
  Other Names: TLI
Drug: Rituximab — Rituximab 375 mg/m2 administered as an intravenous (IV) infusion once weekly for 4 doses.
  Other Names: Rituxan
Drug: Anti-thymoglobulin, rabbit (ATG, rabbit ATG) — Rabbit anti-thymoglobulin (ATG) administered from Day -11 through Day -7 (5 doses) at 1.5 mg/kg/day, for a total dose of 7.5 mg/kg.
Drug: Cyclosporine — Cyclosporine (CSP) administered orally at 6.25 mg/kg twice-a-day (BID) from Day -3 until through Day +56 post-peripheral blood progenitor cell (PBPC) infusion. Dose may be adjusted to maintain a therapeutic level of cyclosporine, or in response to renal insufficiency. If at Day +56, chimerism assessment demonstrates > 40% donor cells in the CD3+ lineage, and the patient is without evidence of GvHD, then cyclosporine taper will begin (6% reduction per week).
  Other Names: CSP; Sandimmune
Drug: Mycophenylate mofetil — Mycophenylate mofetil (MMF) will be administered at 15 mg/kg po Day 0, at 5 to 10 hours after mobilized PBPC infusion is complete
  Other Names: MMF; CellCept
Drug: Filgrastim — Filgrastim provided as needed for neutrophil support
  Other Names: G-CSF; Granulocyte-colony stimulating factor; Neupogen
Drug: Granisetron — Granisetron administered as an anti-nausea agent (anti-emetic) at 1 mg orally 30 to 60 minutes before TLI
  Other Names: Sancuso
Drug: Solumedrol — Solumedrol, an anti-inflammatory glucocorticoid containing methylprednisolone sodium succinate, administered at 1 mg/kg as a premedication for anti-thymoglobulin (ATG)
  Other Names: Medrol; Depo-Medrol; A-Methapred
Drug: Acetaminophen — Acetaminophen administered orally at 650 mg 1 hour prior to infusion of PBPC
  Other Names: Tylenol
Drug: Diphenhydramine — Diphenhydramine administered by intravenous infusion at 50 mg 1 hour prior to infusion of PBPC
  Other Names: Benadryl
Drug: Hydrocortisone — Hydrocortisone administered by intravenous infusion at 100 mg 1 hour prior to infusion of PBPC
  Other Names: Westcort

SUMMARY:
To determine if rituximab administered after allogeneic transplantation decreases the incidence of chronic graft-vs-host disease (cGvHD)

DETAILED DESCRIPTION:
To test if prophylactic anti-B-cell therapy (weekly rituximab) given within 60 to 90 days after allogeneic transplantation will decrease allogeneic donor B-cell immunity and possibly the incidence of chronic graft-vs-host disease (cGvHD).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Between 18 and 76 years of age
* Chronic lymphocytic leukemia (CLL):

  * Unmutated IgG VH gene status
  * Mutated IgG VH genes (> 2% nucleotide change compared to somatic sequence)
  * Complete remission benefit most from allogeneic hematopoietic stem cell transplant (HSCT).

(Physicians will be encouraged to provide aggressive chemotherapy prior to nonmyeloablative transplantation.)

* Mantle cell lymphoma (MCL): Transplant physicians believe subject would benefit from allogeneic HSCT.
* Adequate renal (Cr < 2.4 mg/dL) and hepatic (Bilirubin < 3.0 mg/dL, Aspartate aminotransferase (AST) < 100 IU) function.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* All subjects must provide written informed consent

Donor Inclusion Criteria:

* Genotypically or phenotypically human leukocyte antigen (HLA)-identical.
* Age < 76 unless cleared by institutional PI
* Capable of giving written, informed consent.
* Must consent to peripheral blood stem cell (PBSC) mobilization with G-CSF and apheresis

Recipient Exclusion Criteria:

* Recipient has a 9 of 10 or 10 of 10 HLA identical donor (high resolution molecular genotyping at HLA A, B, C and DrB1, and DQ)
* Pregnancy
* Lactating
* Serious uncontrolled infection
* HIV seropositivity
* Hepatitis B or C seropositivity
* Cardiac function: ejection fraction < 40% or uncontrolled cardiac failure
* Pulmonary: Diffusing capacity - carbon monoxide (DLCO) < 50% predicted
* Liver function abnormalities: elevation of bilirubin to ≥ 3 mg/dL and/or AST > 100
* Renal: creatinine > 2.4
* Karnofsky performance score ≤ 60%
* Patients with poorly controlled hypertension (systolic blood pressure > 150 or diastolic blood pressure > 90 repeatedly).
* Known life-threatening hypersensitivity to rituximab or other anti-B cell antibodies.
* Inability to comply with the allogeneic transplant treatment.
* Uncontrolled central nervous system (CNS) involvement with disease

Donor Exclusion Criteria:

* Identical twin to subject
* Contra-indication to subcutaneous G-CSF at a dose of 16 mg/kg/d for 5 consecutive days
* Serious medical or psychological illness
* Prior malignancy within the preceding five years, with the exception of non-melanoma skin cancers.
* HIV seropositivity

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Result] Arai S, Sahaf B, Narasimhan B, Chen GL, Jones CD, Lowsky R, Shizuru JA, Johnston LJ, Laport GG, Weng WK, Benjamin JE, Schaenman J, Brown J, Ramirez J, Zehnder JL, Negrin RS, Miklos DB. Prophylactic rituximab after allogeneic transplantation decreases B-cell alloimmunity with low chronic GVHD incidence. Blood. 2012 Jun 21;119(25):6145-54. doi: 10.1182/blood-2011-12-395970. Epub 2012 May 4. PMID 22563089

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Rituximab: Participants to receive total lymphoid irradiation + anti-thymoglobulin (TLI + ATG) then nonmyeloablative allogeneic stem cell transplantation, with prophylactic rituximab
Period: Overall Study
Arm/Group | Prophylactic Rituximab
Started | 36
Completed | 33
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by subject (before treatment) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prophylactic Rituximab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 57 [31 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 3
Patient Disease characteristics [Number; unit: participants]
  CLL- Chronic Lymphocytic Leukemia | 22
  MCL- Mantle Cell lymphoma | 13
  unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Chronic Graft-vs-Host Disease (cGvHD)
Description: The cumulative percentage of participants who develop chronic graft-vs-host disease (cGvHD). Chronic cGvHD was defined as at least one instance of a clinically-accepted marker for cGvHD (see Filipovich, et al. Biology of Blood and Marrow Transplantation. 2005;11:945-955)
Time Frame: 4 years
Population: 35 total participants were analyzed. No data is available for the withdrawn participant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Rituximab
Number analyzed (Participants) | 35
percentage of participants | 20 [6 to 34]

2. Secondary Outcome: Incidence of Relapse
Description: Subjects who Relapsed following after Allogeneic HSCT
Time Frame: 4 years
Population: 35 total participants were analyzed. No data is available for the withdrawn participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Rituximab
Number analyzed (Participants) | 35
Participants | 18
Statistical Analysis 1: Comparison: Prophylactic Rituximab; Test type: Superiority or Other; p = .07, Log Rank

3. Secondary Outcome: Mortality
Description: Number of participants who died within 100 days and within 1 year, non-relapse and associated with relapse.
Time Frame: Day 100 and 1 year
Population: 35 total participants were analyzed. No data is available for the withdrawn participant.
Measure: Number; unit: Participants
Arm/Group | Prophylactic Rituximab
Number analyzed (Participants) | 35
Participants
  Mortality within 100 days, all causes | 0
  Nonrelapse mortality within 1 year | 1
  Relapse + mortality within 1 year | 2

4. Secondary Outcome: Overall Survival
Time Frame: 4 years
Population: 35 total participants were analyzed. No data is available for the withdrawn participant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants by disease
Groups:
- Prophylactic Rituximab (CLL Patients): CLL participants to receive total lymphoid irradiation + anti-thymoglobulin (TLI + ATG) then nonmyeloablative allogeneic stem cell transplantation, with prophylactic rituximab
- Prophylactic Rituximab (MCL Patients): MCL participants to receive total lymphoid irradiation + anti-thymoglobulin (TLI + ATG) then nonmyeloablative allogeneic stem cell transplantation, with prophylactic rituximab
Arm/Group | Prophylactic Rituximab (CLL Patients) | Prophylactic Rituximab (MCL Patients)
Number analyzed (Participants) | 22 | 13
Percentage of participants by disease | 73 [57 to 94] | 69 [48 to 99]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Prophylactic Rituximab
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Rituximab (N=35)
Flu-like symptom - Headache (General disorders) | 1 (1)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1 (1)
Acute Graft vs Host Disease (Gastrointestinal disorders) | 1 (1) — Affecting skin, liver and GI tract
Graft vs Host Disease (Blood and lymphatic system disorders) | 1 (1) — Affecting skin, liver, kidney
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Rituximab (N=35)
Flu-like symptoms (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No